CLINICAL TRIAL: NCT07144995
Title: Adjusted Indirect Treatment Comparison of Fruquintinib-based Therapy Versus Standard Care in Advanced Gastric/Gastroesophageal Junction Adenocarcinoma: A MAIC Analysis.
Brief Title: MAIC of Fruquintinib Plus Paclitaxel Versus Ramucirumab Plus Paclitaxel in Advanced G/GEJ Adenocarcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Feng Wang, Professor, Sun Yat-sen University
Other Study IDs: HMPL-013-FLAG-G118
Record Dates: First submitted 2025-08-05; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Advanced Gastric Cancer; Gastroesophageal Junction Adenocarcinoma; Fruquintinib; Ramucirumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fruquintinib + paclitaxel: Group 1: Fruquintinib + Paclitaxel (IPD)
  Interventions: Drug: Fruquintinib+Paclitaxel
- Ramucirumab + paclitaxel: Group 2: Control Therapy (AgD from RAINBOW-Asia)
  Interventions: Drug: Ramucirumab+Paclitaxel

INTERVENTIONS:
Drug: Fruquintinib+Paclitaxel — (using IPD from the FRUTIGA trial, n=703) Fruquintinib：subjects received Fruquintinib orally, once daily for 3 wks on/ 1 wk off Paclitaxel：Paclitaxel 80mg/㎡ at day 1,8,15 of 4-week cycle.
  Other Names: HMPL-013+paclitaxel
  Groups: Fruquintinib + paclitaxel
Drug: Ramucirumab+Paclitaxel — (using published AgD from RAINBOW-Asia, n=440) Ramucirumab：8 milligrams/kilogram (mg/kg) intravenous (IV) infusion on Days 1 and 15 of every 4-week cycle Paclitaxel ：Paclitaxel 80mg/㎡ at day 1,8,15 of 4-week cycle.
  Other Names: LY3009806 +paclitaxel
  Groups: Ramucirumab + paclitaxel

SUMMARY:
This anchored matching-adjusted indirect comparison (MAIC) evaluates the relative efficacy of fruquintinib-paclitaxel (using IPD from the FRUTIGA trial, n=703) versus ramucirumab-paclitaxel (using published AgD from RAINBOW-Asia, n=440) in advanced gastric/GEJ adenocarcinoma. Baseline characteristics are adjusted via entropy balancing weights. Primary endpoint is progression-free survival (PFS) analyzed by Bucher method; secondary endpoints include overall survival (OS) and objective response rate (ORR). Sensitivity analyses comprise restricted mean survival time (RMST) analysis and simulated treatment comparison (STC).

DETAILED DESCRIPTION:
This retrospective MAIC analysis employs individual patient data (IPD) from the FRUTIGA trial (fruquintinib arm) and published aggregate data (AgD) from RAINBOW-Asia (ramucirumab arm), with placebo as the common anchor. Pseudo individual participant data (Pseudo-IPD) for the RAINBOW-Asia trial were reconstructed from published Kaplan-Meier curves using the Guyot algorithm (2012).

•Weighting Methodology: Seven prognostic factors balanced: age <65, male sex, ECOG 0, GEJ primary, peritoneal metastases, metastatic sites, prior doublet chemotherapy Optimization via BFGS algorithm (convergence tolerance 1e-6) Effective sample size (ESS) retention: > 50%

•Statistical Analysis: Primary: Adjusted PFS hazard ratio (HR) using Bucher method with 95% bootstrap CI (100 iterations) Secondary: Weighted Cox models for OS; logistic regression for ORR/DCR Sensitivity: Simulated Treatment Comparison (STC) and covariate threshold analyses

•Sensitivity Analyses: RMST analyses were conducted as supportive evidence alongside primary Cox models for time-to-event endpoints violating proportional hazards assumptions.

Restricted mean survival time (RMST) Simulated Treatment Comparison (STC) Bootstrap confidence intervals (100 iterations)

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed gastric/GEJ adenocarcinoma
* Advanced or metastatic disease
* ECOG 0-1
* Received either fruquintinib + paclitaxel or reference regimen
* Available baseline characteristics for matching variables

Exclusion Criteria:

* Missing key outcome data
* Incomplete baseline characteristics for >2 matching variables
* Prior fruquintinib exposure (control arm only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective MAIC analysis employs individual patient data (IPD) from the FRUTIGA trial (fruquintinib arm) and published aggregate data (AgD) from RAINBOW-Asia (ramucirumab arm), with placebo as the common anchor.
Sampling Method: Non-Probability Sample
Enrollment: 1143 (Estimated)
Dates: Start 2025-09-05 (Estimated); Primary Completion 2026-08-05 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | about 3 years
  Time from randomization to progression/death, assessed via weighted Cox model

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | about 3 years
  CR+PR per RECIST 1.1, compared via weighted logistic regression
Disease Control Rate (DCR) | about 3 years
  CR+PR+SD≥6 weeks, analyzed via weighted proportions
Overall Survival (OS) | about 3 years
  Time from randomization to death, analyzed using weighted Kaplan-Meier
PFS by ECOG, metastasis burden, primary site, etc | about 3 years
  To examine the associations between subgroup factors (including ECOG, metastasis burden, primary site, etc) and Progression-Free Survival (PFS).
OS by ECOG, metastasis burden, primary site, etc | about 3 years
  To examine the associations between subgroup factors (including ECOG, metastasis burden, primary site, etc) and Overall Survival (OS).

OTHER OUTCOMES:
Sensitivity Analyses：Progression-Free Survival (PFS) | about 3 years
  Simulated Treatment Comparison (STC), Bootstrap confidence intervals (100 iterations)

CONTACTS AND LOCATIONS:
Overall Officials: Feng Wang, Principal Investigator — Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: Yes
This study utilizes aggregated data from published literature and de-identified IPD authorized by Hutchison Medipharma Limited. Secondary analysis generated by our team will be shared.
Supporting Information: SAP
Time Frame: Within 6 months after main publication.
Access Criteria: Secondary analysis generated by our team require approval by an independent review committee and a signed data use agreement.
URL: https://www.clinicalstudydatarequest.com

DOCUMENTS (1):
  • Study Protocol (2025-08-01): https://cdn.clinicaltrials.gov/large-docs/95/NCT07144995/Prot_000.pdf